CLINICAL TRIAL: NCT07256314
Title: Investigating the Effects of Diet and Gut Microecology on Bone Health in Gannan Tibetan Elementary School Students
Brief Title: Linking Dietary Nutrition, Dietary Patterns, Gut Microbiota, and Bone Density: A Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: Jianhua Ma (Other)
Responsible Party: Sponsor-Investigator, Jianhua Ma, Lecturer, LanZhou University
Organization: LanZhou University (Other)
Other Study IDs: IRB23082901
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Bone Density; Gut Microbiomes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Faecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Good Bone Density group and normal bone density group
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No Intervention

SUMMARY:
The study aims to understand the current situation of bone health in the Gannan Tibetan primary school student population, to explore the relationship between nutrition, intestinal microorganisms and bone health, to analyze the main factors affecting bone health from the perspective of nutrition and intestinal microecology, and to provide theoretical basis for the promotion and improvement of bone health in Tibetan primary school students.

ELIGIBILITY:
Inclusion Criteria:

* Tibetan primary school students currently enrolled in schools in Gannan Tibetan Autonomous Prefecture;

Willing to participate and able to cooperate in completing bone density measurements;

Additional inclusion criteria: Subjects who are 9 years old or older and agree to participate in dietary surveys and fecal sampling.

Exclusion Criteria:Use of corticosteroid medications within the past year;

Suffering from skeletal system diseases, metabolic disorders, or endocrine diseases;

Additional exclusion criteria: Subjects who have used antibiotics in the past three months and are undergoing fecal sampling.

-

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study is based on a cross-sectional design. Two schools were selected: one rural primary school in Xiahe County, Gannan Tibetan Autonomous Prefecture, and one urban primary school in Hezuo City, Gansu Province. Within the selected schools, a stratified random cluster sampling method was used to randomly select one class from each grade as the study subjects.
Sampling Method: Probability Sample
Enrollment: 431 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Dietary Characteristics | Day 1
  Dietary data were collected using a food frequency questionnaire (FFQ) to analyze dietary patterns and nutrient intake.
Bone density test | Day1
  In this study, a peripheral dual-energy X-ray absorptiometry (EXA-PRESTO) was used to measure the bone density of the non-dominant forearm of the subjects.
Fecal sample microbiological testing and analysis | Day 1
  This study entrusted Tianhao Gene Technology Co., Ltd. to perform the intestinal microbiome Accu16STM (16S rRNA absolute quantitative sequencing). The main research processes include DNA extraction, PCR amplification, library construction, and sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Lanzhou university, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No